CLINICAL TRIAL: NCT04401865
Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-Linking in Eyes With Corneal Thinning Conditions
Brief Title: Safety and Effectiveness of the PXL-Platinum 330 System
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Eye Consultants/Cornea Consultants of Colorado (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PXL-330
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Corneal Ectasia; Keratoconus; Pellucid Marginal Corneal Degeneration
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Pulsed, Accelerated (Experimental): 5 mW, 10 sec on, 10 sec off, 24 minutes of illumination Intervention: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
- Conventional (Active Comparator): 4 mW, 10 sec on, 10 sec off, 30 minutes of illumination Intervention: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution

INTERVENTIONS:
Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution — Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea
  Other Names: Corneal cross-linking

SUMMARY:
To evaluate the safety and effectiveness of the PXL Platinum 330 system for performing corneal cross-linking (CXL) for the treatment of ectatic disorders.

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, intraocular pressure, and pachymetry.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of keratoconus, forme fruste keratoconus, post-LASIK ectasia, pellucid marginal degeneration, forme fruste pellucid marginal degeneration, history of radial keratotomy with fluctuating vision, Terrien's marginal degeneration.
2. Must have provided informed consent, documented it in writing, and have been given a copy of the signed informed consent form.
3. Must be willing and able to return for scheduled treatment and follow-up examinations for the duration of the study.
4. Must be at least 8 years of age.
5. Non-consenting/impaired individuals with a LAR's signature

Exclusion Criteria:

1. Corneal thickness < 300 microns measured by ultrasound or Pentacam.
2. Contraindications or sensitivities to any study medications or their components.
3. Pregnancy or breastfeeding.
4. Any history of Herpes simplex corneal disease in an eye to be treated.
5. Nystagmus or any other condition that would, in the judgement of the investigator, prevent a steady gaze during the treatment.
6. Inability to cooperate with diagnostic tests.
7. Current enrollment in another ophthalmic clinical trial.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Corrected distance visual acuity | 6 months
  Change in corrected distance visual acuity (CDVA) at the last required study visit (6 months post-op), compared to baseline.

SECONDARY OUTCOMES:
Uncorrected visual acuity | 6 months
  Change in UCVA at 6 months, compared to baseline.
Keratometry | 12 months
  Change in Kmax, compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: S. Lance Forstot, M.D., Principal Investigator — Colorado Eye Consultants/Corneal Consultants of Colorado
Locations (3):
- United States (3):
  - Colorado Eye Consultants/Corneal Consultants of Colorado, Littleton, Colorado
  - Chicago Cornea Consultants, Ltd., Highland Park, Illinois
  - Cleveland Eye Clinic, Brecksville, Ohio

IPD SHARING:
Plan to Share IPD: No